CLINICAL TRIAL: NCT00075049
Title: Dbl-Blind, Rand Phase 1/2a Human Challenge Study, to Eval Safety, Reactogenicity, Immunogenicity and Preliminary Efficacy After Sporozoite Challenge/Rechallenge of Vaccines Containing RTS,S
Brief Title: Safety and Efficacy Study of RTS,S AS02A/AS01B Vaccine to Prevent Malaria
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: GlaxoSmithKline (Industry); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: WRAIR 1032; HSRRB A-12227; 257049/027
Record Dates: First submitted 2003-12-31; First posted 2004-01-01 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Malaria
Keywords: malaria
MeSH Terms: conditions — Malaria | interventions — AS01B adjuvant

INTERVENTIONS:
Biological: RTS,S with AS02A/AS01B adjuvant

SUMMARY:
This is a double blinded study where 2 test vaccines will be evaluated to see if they protect persons who have never had malaria against malaria infection when bitten by mosquitoes.

ELIGIBILITY:
Inclusion Criteria:

* Be in good general health
* Be able to participate for 4-15 months

Exclusion Criteria:

* Pregnant or planning pregnancy
* History of malaria or exposure to malaria in past 12 months
* Received an investigational malaria vaccine
* Past history of allergic reaction to previous immunization
* Positive blood tests for HIV and specific types of hepatitis

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104
Dates: Start 2003-12; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
To assess the safety and reactogenicity of the candidate vaccine

SECONDARY OUTCOMES:
To assess the humoral immune response to the candidate vaccine
To assess the efficacy of the candidate vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Kent Kester, MD, Principal Investigator — Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- Walter Reed Army Institute of Research, Silver Spring, Maryland, United States

REFERENCES:
- [Result] Stewart VA, McGrath SM, Walsh DS, Davis S, Hess AS, Ware LA, Kester KE, Cummings JF, Burge JR, Voss G, Delchambre M, Garcon N, Tang DB, Cohen JD, Heppner DG Jr. Pre-clinical evaluation of new adjuvant formulations to improve the immunogenicity of the malaria vaccine RTS,S/AS02A. Vaccine. 2006 Oct 30;24(42-43):6483-92. doi: 10.1016/j.vaccine.2006.06.033. Epub 2006 Jul 3. PMID 16904798
- [Derived] Kurtovic L, Atre T, Feng G, Wines BD, Chan JA, Boyle MJ, Drew DR, Hogarth PM, Fowkes FJI, Bergmann-Leitner ES, Beeson JG. Multifunctional Antibodies Are Induced by the RTS,S Malaria Vaccine and Associated With Protection in a Phase 1/2a Trial. J Infect Dis. 2021 Oct 13;224(7):1128-1138. doi: 10.1093/infdis/jiaa144. PMID 32236404
- [Derived] Kester KE, Cummings JF, Ofori-Anyinam O, Ockenhouse CF, Krzych U, Moris P, Schwenk R, Nielsen RA, Debebe Z, Pinelis E, Juompan L, Williams J, Dowler M, Stewart VA, Wirtz RA, Dubois MC, Lievens M, Cohen J, Ballou WR, Heppner DG Jr; RTS,S Vaccine Evaluation Group. Randomized, double-blind, phase 2a trial of falciparum malaria vaccines RTS,S/AS01B and RTS,S/AS02A in malaria-naive adults: safety, efficacy, and immunologic associates of protection. J Infect Dis. 2009 Aug 1;200(3):337-46. doi: 10.1086/600120. PMID 19569965